CLINICAL TRIAL: NCT04398303
Title: A Phase 1/2 Randomized, Placebo-Controlled Trial of ACT-20 in Patients With Severe COVID-19 Pneumonia
Brief Title: ACT-20 in Patients With Severe COVID-19 Pneumonia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aspire Health Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHS 20-03
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: COVID-19 Pneumonia
Keywords: Stem cells; Pneumonia; COVID; COVID-19; Coronavirus; SARS-CoV-2
MeSH Terms: conditions — Pneumonia; COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ACT-20-MSC in ACT-20-CM (Experimental): Conventional treatment plus ACT-20-MSC in ACT-20-CM administered intravenously
  Interventions: Biological: ACT-20-MSC
- ACT-20-CM (Experimental): Conventional treatment plus ACT-20-CM administered intravenously
  Interventions: Biological: ACT-20-CM
- Placebo (Placebo Comparator): Conventional treatment plus placebo (MEM-α) administered intravenously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ACT-20-MSC — 1 million cells / kg body weight in 100 ml in conditioned media
  Arms: ACT-20-MSC in ACT-20-CM
Biological: ACT-20-CM — 100 ml of conditioned media only
  Arms: ACT-20-CM
Biological: Placebo — 100 ml of MEM-α
  Arms: Placebo

SUMMARY:
The primary objective of this study is determine the safety and efficacy of ACT-20-MSC (allogenic human umbilical derived mesenchymal stem cells) and ACT-20-CM (allogenic human umbilical derived mesenchymal stem cells in conditioned media) in patients with moderate to severe COVID-19 pneumonia.

DETAILED DESCRIPTION:
This study will assess the safety and efficacy of ACT-20-MSC and ACT-20-CM administered intravenously to subjects with moderate to severe COVID-19 related pneumonia in two parts.

Part 1 is an open-label study of 10 subjects, 5 with moderate COVID-19 pneumonia and 5 with severe COVID-19 pneumonia. Of these 10 subjects, 5 will receive ACT-20-CM and 5 will receive ACT-20-MSC resuspended in ACT-20-CM.

Part 2 is a randomized, blinded, placebo-controlled study of 60 patients, 30 with moderate COVID-19 pneumonia and 30 with severe COVID-19 pneumonia. Randomization will be 1:1:1 ACT-20-MSC in ACT-20-CM, ACT-20-CM or placebo. The placebo is MEM-α, a widely used sterile culture media that contains non-essential amino acids, nucleosides, vitamins, glucose, sodium pyruvate and lipoic acid.

Subjects treated at each investigative site will provide written informed consent prior to the conduct of any study-related procedures. Thereafter, they will be screened and those meeting the inclusion/exclusion criteria will be enrolled into the trial and undergo all the study procedures including the intravenous administration of the investigational medical product (IMP = ACT-20-MSC in ACT-20-CM or ACT-20-CM) or placebo. The IMP will be administered in addition to any standard of care treatment the subject is receiving.

Subjects will be assessed daily while in hospital. Following discharge from hospital, subjects will be following for an additional three month period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age 18 to 85, inclusive
2. Confirmed positive test for COVID-19 by standard reverse transcriptase polymerase chain reaction (RT-PCR) assay or equivalent
3. On mechanical ventilation (n=35), or high-flow O2 support (n=35) and:

   1. Disease severity level of "moderate" (PaO2/FiO2 of 100-200) (n=35), or "severe" (PaO2/FiO2 < 100) (n=35) as established using the Berlin Criteria for ARDS (Barbas, Isola & Caser, 2014; Baron & Levy, 2016).
   2. Positive end-expiratory airway pressure (PEEP) ≥ 5 cmH2O
   3. Oxygen saturation ≤ 93%
4. Non-cardiogenic bilateral pulmonary edema on frontal chest radiograph that cannot be explained by effusion, collapsed lung or lung nodule
5. Able to understand and provide voluntary informed consent

Exclusion Criteria:

1. Unable to understand and provide voluntary informed consent
2. Current infection with HIV-1, HIV-2, Hepatitis B, Hepatitis C or HTLV
3. History of malignancy, other than non-melanoma skin cancer or non-metastatic prostate cancer
4. Currently receiving extracorporeal life support or high-frequency oscillatory ventilation
5. Weight > 150 kg
6. Current severe chronic respiratory disease, as demonstrated by:

   1. PaCO2 > 50 mm Hg, or
   2. history of use of home oxygen
7. Major trauma within the past 7 days
8. Lung transplant recipient
9. WHO Class III or IV pulmonary hypertension
10. Documented deep vein thrombosis or pulmonary embolism within the past 3 months
11. Currently pregnant or lactating
12. Currently participating in another clinical trial, or participation in another clinical trial within 30 days of enrollment
13. Hypersensitivity to Dextran-40 or Dimethyl Sulfoxide (DMSO)
14. Current pharmacotherapy using hydroxychloroquine or Interleukin-6 inhibitors
15. History of CVA or MI within 180 days of study enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Mortality at day 30 | 30 days post treatment

SECONDARY OUTCOMES:
Ventilated Subjects - Ventilator Free Days | 28 days post treatment
  Number of ventilator-free days
Ventilated Subjects - Improvement in Ventilator Settings | 28 days post treatment, or until off of ventilator
  Improvement in ventilator settings: Minute ventilation, PEEP, FiO2
High-Flow O2 Support Subjects - Step-Down O2 Therapy | 30 days post treatment, or until off of high-flow O2 support
  Days of step-down O2 therapy as evidenced by: improvement in required volume, change to nasal cannula or face mask delivery or improvement in required concentration.
High Flow O2 Support Subjects - Respiration Rate | 30 days post treatment, or until off of high-flow O2 support
  Respiration Rate < 30 for > 24 hours.
Both Ventilated and High-Flow O2 Support Subjects - ICU-Free Days | 30 days post treatment, or until off of ventilator or high-flow O2 support
  Number of ICU-free days
Both Ventilated and High-Flow O2 Support Subjects - Pulmonary Function Improvement | 30 days post treatment, or until off of ventilator or high-flow O2 support
  Improvement in pulmonary function as evidenced by A-A oxygen gradient, O2 saturation
Both Ventilated and High-Flow O2 Support Subjects - Increased Berlin Score | 30 days post treatment, or until off of ventilator or high-flow O2 support
  Increased Berlin Criteria score > 24 hours

REFERENCES:
- See also: Related Info — http://aspire2cure.com